CLINICAL TRIAL: NCT03359317
Title: Jogging in the Change of Osteoporosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Shenzhen Sun Yat-sen Cardiovascular Hospital (Other); Wujin People's Hospital (Other); Chongqing Zhongshan Hospital (Other Government)
Responsible Party: Principal Investigator, Zhang Yichong, Department of orthopaedics and trauma, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKUPH-JGO
Record Dates: First submitted 2017-11-26; First posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Bone Diseases
MeSH Terms: conditions — Osteoporosis; Bone Diseases | interventions — Jogging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- jogging (Experimental): At least 5 times/week
  Interventions: Behavioral: jogging

INTERVENTIONS:
Behavioral: jogging — Jogging as instructed for 1 year

SUMMARY:
To test the changes in osteoarthritis according to the X-rays, and changes in bone quality before and 1 or more years after beginning the jogging

DETAILED DESCRIPTION:
Patients in this research are given an entry Bone Densitometry（DEXA）scan and are required to advance from 3-minute jogging a day to 10-minute level in daily practice for 1 year as instructed. After 1 year, subsequent DEXA scans are recorded. Interested participants are also encouraged to have hip and spine X-rays, and bone quality studies on study entry and two years later. Actual subject participation, intercurrent illnesses, fractures and changes in medication are self-monitored. Results are calculated by change in bone mineral density in the lumbar spine, hips and femurs by the DEXA scan in the study. Dose-response relationships between the amount of jogging and bone mineral density are sought. Jogging-related fractures and other adverse effects are also noted.

ELIGIBILITY:
Inclusion Criteria:

Past DEXA scan and, all within 6 months of study entry, DEXA scan and normal values for: Metabolic panel, TSH, PTH, ESR (or CRP), Vitamin D 25 hydroxy, Vitamin D 1,25 dihydroxy, Urine NTX

Exclusion Criteria:

Known metabolic bone disease such as osteogenesis imperfecta, current treatment with steroids, chemotherapy, or currently healing fractures of lumbar spine, hips or femurs, severe heart disease

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-02-20 (Estimated); Primary Completion 2019-01-30 (Estimated); Study Completion 2019-01-30 (Estimated)

PRIMARY OUTCOMES:
DEXA T-score | 1 year
  Bone mineral density change in spine, hip and femur after 1 year of jogging

SECONDARY OUTCOMES:
Number of fractures | 1 year
  Number of fractures occurring while in study

CONTACTS AND LOCATIONS:
Overall Officials: Peixun Zhang, MD, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No